CLINICAL TRIAL: NCT01114854
Title: A Conversion Study to Determine the Relative Bioavailability of TPM MR vs TPM IR in Subjects With Epilepsy
Brief Title: A Conversion Study of Immediate Release (IR) and Modified Release (MR) Forms of Topiramate (TPM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 538P108
Record Dates: First submitted 2010-04-28; First posted 2010-05-03 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Topiramate

STUDY DESIGN:
Masking Description: It was a open-label study
Oversight: Data Monitoring Committee: No

ARMS (1):
- Topiramate IR followed by Topiramate ER (Other): Dosing with IR followed by dosing with ER
  Interventions: Drug: Topiramate IR; Drug: Topiramate ER

INTERVENTIONS:
Drug: Topiramate IR
  Other Names: Topamax®
Drug: Topiramate ER
  Other Names: SPN-538T

SUMMARY:
This multi-center, two-treatment study compares the pharmacokinetic profiles of Immediate Release (IR) and Modified Release (MR) formulations of Topiramate (TPM) in patients with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female patients with epilepsy on stable doses of topiramate.
2. Able to voluntarily provide written informed consent to participate in the study.
3. Use of an effective form of birth control if of child-bearing potential.

Exclusion Criteria:

1. Diagnosis of status epilepticus, non-epileptic seizures, or any progressive CNS disease.
2. Recent or recurrent suicidal thoughts or ideation.
3. Clinically significant medical condition that may affect the safety of the subject.
4. Females who are pregnant or lactating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
relative bioavailability at steady-state of TPM MR and TPM IR, as determined by TPM levels in plasma | 2 weeks

SECONDARY OUTCOMES:
relative bioavailability of TPM MR immediately following switch from TPM IR, as determined by TPM levels in plasma | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Baroldi, MD, PhD, Study Director — Supernus Pharmaceuticals, Inc.
Locations (9):
- United States (9):
  - Kyle Patrick, Phoenix, Arizona
  - Victor Biton, Little Rock, Arkansas
  - Mohammed Bari, National City, California
  - Dr. Segal, Fort Lauderdale, Florida
  - Dr. Sackellares, Gainesville, Florida
  - James Kiely, Atlanta, Georgia
  - Bassem El-Nabbout, Wichita, Kansas
  - Dr. Chumley, Lexington, Kentucky
  - Dr. Fisher, Oklahoma City, Oklahoma